CLINICAL TRIAL: NCT06695754
Title: A Systematic Review and Meta-Analysis to Compare the Effectiveness of Manual and Automatic Colonic Massage Interventions in Patients With Chronic Constipation.
Brief Title: Comparing Manual and Automatic Colonic Massage for Chronic Constipation.
Acronym: COMACOMACC
Status: Completed | Type: Observational
Sponsor: usMIMA S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: MOW_07_2024
Record Dates: First submitted 2024-11-13; First posted 2024-11-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Constipation
Keywords: manual massage; automatic massage; colonic massage; intermittent colonic exoperistalsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Manual massage <90% over colon: Patients received a manual massage or treatment that reachs the ascending and descending colon for less than 90% of the total time of the treatment duration
- Manual massage >90% over colon: Patients received a manual massage or treatment that reachs the ascending and descending colon for 90% or more of the total time of treatment duration
- Automatic massage: Patients received a massage or treatment delivered with a medical device, that reachs the ascending and descending colon for 90% or more of the total time of treatment duration

SUMMARY:
The aim of this study is to do a systematic review and metanalysis of the scientific literature to compare the effectiveness of the manual vs the automatic colonic massage intervention in patients with chronic constipation.

DETAILED DESCRIPTION:
Retrieval Strategy

* Computer retrieval of clinical literature on abdominal massage for constipation published between 1990 and December 2024 will be conducted in:

  * NCBI PubMed.
  * Research Gate.
  * Google Scholar.
  * Ovid.
* English retrieval terms included: colon, abdominal, constipation, bowel function, transit time, massage, and device.
* A cross-retrieval will be conducted to screen the literature that met the inclusion criteria.

Literature screening and data extraction

* The literature search will be independently performed by two researchers.
* Identified studies will be imported into EndNote×9 and Mendeley for organization.
* Articles will be evaluated based on predefined inclusion and exclusion criteria.
* Duplicates from various databases will be removed.
* Clearly irrelevant articles will be excluded based on their titles and abstracts.
* Full texts of the remaining studies will be thoroughly reviewed, and those that met the criteria will be included.
* The final dataset will be cross-verified.
* Discrepancies will be resolved through discussion or by involving a third researcher with a PhD for arbitration.
* Extracted data included:

  * First author's name
  * Publication year
  * Study type
  * Sample size
  * Participant gender and age
  * Interventions in both experimental and control groups
  * Treatment duration and frequency
  * Primary and secondary study outcomes
  * Quality assessment of the studies
* Study characteristics, along with the study design, description of interventions (type of colon massage applied), and indices of evaluated results, will be organized using an Excel-based data extraction form.

Quality evaluation

* Quality assessment of the literature will be conducted using the "risk of bias" tool recommended by the Cochrane Handbook for Systematic Reviews (Rob2.0 and Robins-E). These tools evaluate various bias domains, including randomization, deviations from intended interventions, missing data, outcome measurement, and selective reporting. Each domain will be rated as having a high, unclear, or low risk of bias.
* Disagreements between the two researchers regarding the literature's conclusions will be resolved through discussion or by a third researcher.

ELIGIBILITY:
Literature Inclusion Criteria:

* Study type:

  * Clinical studies using abdominal/colon massage to treat constipation.
  * Articles published between 1990 and till the day of literature search with original work (experimental and quasi-experimental ) or dealing with the application of colon massage to gastrointestinal function.
* Study subjects:

  * Patients with constipation.
  * Individuals of any gender, age and ethnicity.
* Interventions:

  - Manual or automatic colon massage treatment for constipation.
* Outcomes (including at least one of the following):

  * Evacuation frequency.
  * Quality of life parameters.
  * Symptoms of constipation.
  * Use of laxatives or enemas.
  * Adverse events.

Literature Exclusion Criteria:

* No abstract available, reviews, conference abstracts, dissertations, registration documents, clinical experience summary analysis, animal experiments, etc.
* Studies where the treatment was non-colon specific.
* Studies involving invasive treatments.
* Other treatments intended to treat constipation such as surgical interventions, acupuncture, acupoint application, and others considered medicinal alternative therapies.
* Documents written in languages other than in English, German, Spanish, as well as other European languages, including Italian, French, and Portuguese.
* Incorrect or incomplete case data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of any age, gender and etnicity, suffering from chronic constipation
Sampling Method: Non-Probability Sample
Enrollment: 2312 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Quantitative evaluation of manual vs. automatic colon massage for chronic constipation relief | 34 years
  Quantitative comparison of manual and automatic colon massage efficacy in relieving chronic constipation

SECONDARY OUTCOMES:
Evacuation frequency | 34 years
  Number of bowel movementes per week
Quality of life questionnaire in relation to constipation | 34 years
  Semi-Quantitative score derived from standardized qualitative questionnaires evaluating quality of life in relation to chronic constipation.
Adverse events | 34 years
  Any secondary adverse effect directly derived from the treatment, including Serious Adverse Events (SAE)
Aids to evacuation | 34 years
  Use (total number of days in use or total dose per week) of any aid to facilitate evacuation such as laxatives, enemas, digitation....

CONTACTS AND LOCATIONS:
Overall Officials: Immaculada Herrero-Fresneda, PhD, Study Director — usMIMA S.L.; Eugenia Delgado, PhD, Principal Investigator — usMIMA S.L.
Locations (1):
- Usmima S.L., Esplugues de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No